CLINICAL TRIAL: NCT06760936
Title: Pixantrone as Bridging Therapy to Allogenic Transplant or CAR-T Cell Therapy in DLBCL Patients - A Retrospective-prospective Observational Study
Brief Title: Pixantrone as Bridging Therapy to Allogenic Transplant or CAR-T Cell Therapy in DLBCL Patients
Acronym: PIXBRIDGE
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PIXBRIDGE
Record Dates: First submitted 2024-12-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: pixantrone; allogenic transplant; CAR-T therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective/prospective observational multicentric study aimed at describing the effectiveness of pixantrone as bridging therapy to allo-HSCT or CAR-T therapy

DETAILED DESCRIPTION:
The treatment of relapsed/refractory (R/R) diffuse large B-cell lymphomas (DLBCL) presents a challenge to physicians due to the lack of treatment options. Pixantrone is an aza-anthracenedione, which, compared to anthracyclines and anthracenediones, has significantly reduced cardiotoxicity while maintaining good antitumour activity. The applications of pixantrone can be manifold: elderly patients with a second relapse who are unsuitable for transplantation or CAR-T cell therapy, young patients refractory to 2 previous lines of therapy as a bridge to autologous transplantation, bridge to allogeneic transplantation or CAR-T cell therapy, and salvage therapy for relapses after a transplantation or CAR-T approach. In particular, pixantrone could be one of the most suitable agents to link patients to CAR-T cell therapy due to its safety profile and its ability to induce a rapid response in patients sensitive to this agent. However, data in normal clinical practice are still lacking. Hence the need for an Italian multicentre collection to collect as many cases as possible of patients who have received pixantrone as a bridging therapy to allogeneic transplantation or CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory DLBCL who received pixantrone as last line of therapy prior to allo-HSCT or CAR-T cell therapy or patient's whose therapeutic program is treatment with pixantrone prior to allo-HSCT or CAR-T cell therapy.
2. Age ≥ 18 years at enrolment.
3. Written informed consent (if applicable).

Exclusion Criteria:

1) none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic relapse/refractory DLBCL patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of pixantrone as bridging therapy to allo-HSCT or CAR-T therapy. | through study completion, an average of 2 years
  Number of patients able to proceed to transplant/CAR-T

SECONDARY OUTCOMES:
Treatment duration | through study completion, an average of 2 years
  Mean treatment duration (time required to achieve a response sufficient to led the patient to allo-HSCT or CAR-T Therapy)
patient's response to the treatment with pixantrone | through study completion, an average of 2 years
  Overall response rate (proportion of patients achieving a complete remission, partial remission, stable disease or progressive disease) following treatment with pixantrone
type of adverse events (AE) | through study completion, an average of 2 years
  treatment's tolerability
Assessment of OS | through study completion, an average of 2 years
  patient's survival after both pixantrone and allogenic transplant/CAR-T
causes of discontinuation | through study completion, an average of 2 years
  causes of treatment discontinuation
Incidence of adverse events (AE) | through study completion, an average of 2 years
  treatment's tolerability
Incidence serious adverse events (SAE) | through study completion, an average of 2 years
  treatment's tolerability
type of serious adverse events (SAE) | through study completion, an average of 2 years
  treatment's tolerability
PFS (progression free survival) | through study completion, an average of 2 years
  patient's survival after both pixantrone and allogenic transplant/CAR-T
disease free survival (DFS) | through study completion, an average of 2 years
  patient's survival after both pixantrone and allogenic transplant/CAR-T

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No